CLINICAL TRIAL: NCT02970890
Title: Effects of Photobiomodulation Therapy (PBMT) on Acute Pain and Inflammation in Patients Who Underwent Total Hip Arthroplasty
Brief Title: Effects of Photobiomodulation Therapy (PBMT) in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriane Aver Vanin (Other)
Responsible Party: Sponsor-Investigator, Adriane Aver Vanin, MsC, PhD candidate, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 066490
Record Dates: First submitted 2016-11-01; First posted 2016-11-22 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Total Hip Arthroplasty (THA); Phototherapy; Low-level laser therapy; Light-emitting diodes
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Subjects received placebo therapy. The placebo Portable Pain Away™ device was identical to the active device, displayed the same settings and emitted the same sound regardless of the comparator.
  Interventions: Device: Portable Pain Away™
- PBMT group (Active Comparator): Subjects received active photobiomodulation therapy (PBMT). The active Portable Pain Away™ device was identical to the placebo device, displayed the same settings and emitted the same sound.
  Interventions: Device: Portable Pain Away™

INTERVENTIONS:
Device: Portable Pain Away™ — Portable Pain Away™ device (manufactured by Multi Radiance Medical, Solon - OH, USA) - placebo or active phototherapy
  Other Names: Photobiomodulation therapy (PBMT)

SUMMARY:
Osteoarthritis (OA), a chronic degenerative muscle disease characterized by cartilage wear, causes progressive joint deformity and loss of function leading to the indication of total hip arthroplasty (THA), when conservative treatments fail. Surgical trauma leads to pain and induces an immune response. Photobiomodulation therapy (PBMT) has proven effective in tissue repair by modulating the inflammatory process and promoting pain relief. It can therefore be part of the treatment. This study aims to analyze the effect of PMBT on inflammation and pain of patients who underwent total hip arthroplasty. The study consisted of eighteen patients who underwent hip arthroplasty and they received phototherapy in a period from 8 to 12 hours after surgery. We divided the patients into two groups (n=9 each) placebo and effective phototherapy. The patients were evaluated before and after phototherapy with 9 diodes, applied to 5 points along the scar (1 laser 905nm, 4 LEDs 875nm and 4 LEDs 640nm, 40.3J total), by visual analogue scale (VAS) and blood collection for analysis of the levels of the cytokines TNF-α, IL-6 and IL-8.

ELIGIBILITY:
Inclusion Criteria:

- Men and women with clinical diagnosis of OA based on radiological images in the anteroposterior and profile according to Demur classification.

Exclusion Criteria:

- Men and women with other clinical diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of Pain (VAS) | Change from baseline in VAS to immediately after phototherapy
  A visual analogue scale (VAS) of 100 mm was used for the self-rating of the patients pain intensity, with assistance of a blinded researcher. Pain assessments were performed at baseline, immediately after phototherapy irradiation.
Evaluation of Cytokines levels (ELISA immunoenzymatic assay) | Change from baseline in Cytokines levels to immediately after phototherapy
  Cytokine levels (IL-6, IL-8 and TNF-α) in blood samples collected from patients before and after irradiation of phototherapy were evaluated using the Duo Set kit (BD Biosciences) according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beneficência Nossa Senhora do Pari, São Paulo, São Paulo, Brazil